CLINICAL TRIAL: NCT00862875
Title: Effects of Basal Insulin Analogue Detemir on Body Composition, Epicardial Fat and Energy Metabolism
Brief Title: Levemir-Body Composition and Energy Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Novo Nordisk A/S (Industry); McMaster University (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, MD, PhD, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRL-01-2009
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes
Keywords: Insulin initiation; oral therapy failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Glargine; Insulin, Long-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:Insulin detemir (Experimental): Insulin detemir (Levemir® - Novolin® 4 pen)
  Interventions: Drug: Detemir or Glargine
- 2:Insulin Glargin (Active Comparator): Insulin glargine (Lantus® - Solostar®)
  Interventions: Drug: Detemir or Glargine

INTERVENTIONS:
Drug: Detemir or Glargine — Initial dose of 10 units of insulin at bedtime. The insulin dose will be increase by 1 unit per day until fasting plasma glucose (FPG) levels are 5.0 mmol/L.
  Other Names: Detemir; Levemir; Long acting insulin; Bed time insulin; Lantus; basal insulin analogue

SUMMARY:
The objectives is to compare the changes in body composition (primary objective), diabetes parameters, energy expenditure and energy intake between Insulin detemir (Levemir® - Novolin® 4 pen) and insulin glargine (Lantus® - Solostar®) both in combination with Metformin and insulin secretagogues (SU) between baseline and after 6 months of insulin therapy in 80 type 2 diabetic patients failing on oral diabetic agents .

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients who require basal (long-acting) insulin for the control of hyperglycemia according to the opinion of the investigator.
* Inadequate Glucose control: Hemoglobin A1c (HbA1c) percentage in the range of ≥ 7.5 - 12.0%
* Stable body weight for previous 3 months (± 5 kg).
* Structured exercise lower than 4 hours per week.
* Metformin ≥1.5 g/day

Exclusion Criteria:

* Any medical, social or geographic condition, which, in the opinion of the investigator would not allow safe or reliable completion of the protocol.
* Type 1 Diabetes Mellitus
* Previous treatment with insulin (< 6 months prior inclusion). Insulin therapy for less than 6 days at the time of an acute event is acceptable.
* Secondary diabetes mellitus (i.e. steroid induced, Cushing syndrome, chronic pancreatitis, cystic fibrosis, etc.) and maturity-onset diabetes of the young
* Proliferative retinopathy/maculopathy requiring treatment
* Hypoglycemia unawareness or recurrent major hypoglycaemia
* Pregnancy and breast-feeding
* Unstable coronary artery disease
* Heart Failure as defined by class IV according to NYHA classification
* Recent (< 6 months) history of myocardial infarction, stroke or T.I.A, ventricular arrhythmias, or unstable supra-ventricular arrhythmias.
* Renal Insufficiency. Creatinine clearance < 40 ml/min (MDRD formula).
* Acute (< 2 months) or Chronic infectious diseases requiring either hospitalization or antibiotic treatment for more than 2 weeks
* Recent (< 1 year) diagnosis of systemic malignancies except thyroid and skin cancer
* Major psychiatric diseases
* History of drug addiction
* Previous bariatric surgery
* Medication that affects weight such as

  * Systemic corticosteroids (prednisone)
  * Anti-obesity medication (Xenical® or Meridia®)
  * Megace ®
  * Antidepressant medication associated with significant weight impact such as Zyprexa®, Remeron® based on investigator judgment.
  * Growth hormone therapy or testosterone supplementation should be initiated for at least 6 months and at stable dose for 3 months prior to enrolment
  * Medication that affects glycemic control and hypoglycemic unawareness based on investigator judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in total fat mass (in kg) | Baseline and 6 months

SECONDARY OUTCOMES:
Epicardial fat, trunk fat, total fat free mass, weight & waist circumference, HbA1c, fasting glucose, RMR, TEF,PAEE & TEE, energy intake. | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada